CLINICAL TRIAL: NCT02280460
Title: Extracorporeal Membrane Oxygenation(ECMO): Optimization of Its Use
Brief Title: ECMO: Optimization of Its Use
Status: Terminated | Type: Observational
Why Stopped: Study was not able to achieve primary objective and there is no intention to work towards its achievement
Sponsor: Renzo Loyaga Rendon (Other)
Collaborators: Corewell Health West (Other)
Responsible Party: Sponsor-Investigator, Renzo Loyaga Rendon, Medical Director, Cardiovascular Research, Corewell Health West
Organization: Corewell Health West (Other)
Other Study IDs: 2014-194
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Extracorporeal Membrane Oxygenation Complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VA ECMO: Patients who are placed on VA ECMO.
- VV ECMO: Patients who are placed on VV ECMO.

SUMMARY:
To create a local registry for ECMO patients.

DETAILED DESCRIPTION:
To create a local registry of retrospective and prospective patients on ECMO at Spectrum Health, Butterworth campus in order to optimize the use of ECMO therapy and to create algorithms to estimate the prognosis. ECMO patients will be compared to a control group of patients. Patient mortality will be assessed in-house, at 48 hours, 3 months, and 1 year after the start of ECMO therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* requiring ECMO. For the control,Patients without ECMO admited to ICU.

Exclusion Criteria:

* Age<18
* Known prisoner of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Spectrum Health requiring ECMO therarpy. For the control, patients in the Intensive Care Unit at Spectrum Health will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2014-09; Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 year

SECONDARY OUTCOMES:
all cause mortality | 48 hours
In-house mortality | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Loyaga-Rendon, MD,PhD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Zapol WM, Snider MT, Hill JD, Fallat RJ, Bartlett RH, Edmunds LH, Morris AH, Peirce EC 2nd, Thomas AN, Proctor HJ, Drinker PA, Pratt PC, Bagniewski A, Miller RG Jr. Extracorporeal membrane oxygenation in severe acute respiratory failure. A randomized prospective study. JAMA. 1979 Nov 16;242(20):2193-6. doi: 10.1001/jama.242.20.2193. PMID 490805
- [Background] Peek GJ, Mugford M, Tiruvoipati R, Wilson A, Allen E, Thalanany MM, Hibbert CL, Truesdale A, Clemens F, Cooper N, Firmin RK, Elbourne D; CESAR trial collaboration. Efficacy and economic assessment of conventional ventilatory support versus extracorporeal membrane oxygenation for severe adult respiratory failure (CESAR): a multicentre randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1351-63. doi: 10.1016/S0140-6736(09)61069-2. Epub 2009 Sep 15. PMID 19762075